CLINICAL TRIAL: NCT04271020
Title: Urodynamic Feasibility Study (UDS)
Brief Title: Urodynamic Feasibility Study Utilizing the UroLift® System
Acronym: UDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeoTract, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP00009
Record Dates: First submitted 2020-02-04; First posted 2020-02-17 (Actual); Results first posted 2020-05-22 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-05

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- UroLift (Experimental)
  Interventions: Device: UroLift

INTERVENTIONS:
Device: UroLift — The UroLift System is indicated for the treatment of symptoms due to urinary outflow obstruction secondary to benign prostatic hyperplasia (BPH).
  During the procedure, an implant is delivered into the prostatic lobe obstructing the urethra and restricting urine flow. The distal end of the device is used to compress the lobe then the implant is delivered to retain the lobe in position, thereby increasing the urethral opening and reducing the fluid obstruction through the prostatic urethra.

SUMMARY:
UDS evaluates the impact of Prostatic Urethral Lift (PUL) as measured by pressure flow, urodynamic testing (UDS) and an optional UroCuff Testing, an alternative urodynamic test. In addition, standard BPH measures such as symptoms, qualify of life, uroflowmetry, and post void residual will be evaluated at screening and at the follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Male gender
* Diagnosis of symptomatic BPH
* Age ≥ 45 years
* International Prostate Symptom Score (IPSS) ≥ 13
* Peak urine flow rate ≤ 12 ml/sec, voided volume ≥ 125 ml
* Prostate volume ≤ 80 cc per ultrasound

Exclusion Criteria:

* Current urinary retention
* Post void residual (PVR) urine > 250 ml
* Have an obstructive or protruding median lobe of the prostate
* Active urinary tract infection at time of treatment
* Current gross hematuria
* Previous BPH surgical procedure
* Previous pelvic surgery or irradiation
* History of neurogenic or atonic bladder
* Stress urinary incontinence
* Biopsy of the prostate within the past 6 weeks
* Life expectancy estimated to be less than 1 year
* History of prostate or bladder cancer
* Elevated Prostate-Specific Antigen (PSA) without ruling out prostate cancer
* History of compromised renal function or upper tract disease
* Known coagulopathies or subject on anticoagulants or antiplatelets other than aspirin ≤ 100 mg (unless antiplatelets are withheld minimum 3 days prior to procedure)
* Use of the following medications pre-screening (uroflow, questionnaires):

  * Within 4 months of baseline assessment: estrogen, any drug producing androgen suppression, or anabolic steroids
  * Within 3 months of baseline assessment: 5-alpha-reductase inhibitors
  * Within 2 weeks of baseline assessment: alpha-blockers, gonadotropin-releasing hormonal analogs, anticholinergics or cholinergic medication or phenylephrine, pseudoephedrine, or imipramine medications
  * Within 1 week of baseline assessment, unless documented on stable dose for ≥ 6 months: beta blockers, antidepressants, anticonvulsants, and antispasmodics
* Cystolithiasis within the prior 3 months
* History of co-morbidities that would affect having an elective urological procedure including: prostatitis, conditions that preclude the insertion of the UroLift System.
* Other co-morbidities that could impact the study results such as:
* Severe cardiac arrhythmias uncontrolled by medications or pacemaker
* Congestive heart failure New York Heart Assocation (NYHA) III or IV
* History of uncontrolled diabetes mellitus
* Significant respiratory disease in which hospitalization may be required
* Known immunosuppression (i.e. AIDS, post-transplant, undergoing chemotherapy)
* A known allergy to nickel, titanium, or stainless steel
* Unable or unwilling to complete all required questionnaires and follow up assessments
* Unable or unwilling to sign informed consent form
* Currently enrolled in any other investigational clinical research trial that has not completed the primary endpoint.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients must be male. The study is evaluation the population of men diagnosed with benign prostatic hyperplasia.
Enrollment: 12 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Mazzarella, MD, Principal Investigator — Midtown Urology Associates
Locations (1):
- Midtown Urology Associates, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | UroLift
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | UroLift
Number analyzed (Participants) | 12
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 57.44 (6.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Qmax [Mean (Standard Deviation); unit: mL/sec] | 7.0 (2.7)
Pdet @ Qmax [Mean (Standard Deviation); unit: cmH20] — Population: Unable to interpret data from 3 subjects collected at baseline.
  cmH20
    number analyzed (Participants) | 9
    (all) | 79.9 (25.2)
Pdetmax [Mean (Standard Deviation); unit: cmH20] — Population: Unable to interpret data from 3 subjects collected at baseline.
  cmH20
    number analyzed (Participants) | 9
    (all) | 108.9 (34.4)

OUTCOME MEASURES:

1. Primary Outcome: Qmax Assessed Using Urodynamic Testing (Cystometry)
Description: Qmax is the the maximum urinary flow rate measured in ml/s.
Time Frame: 3 Month
Measure: Mean (Standard Deviation); unit: mL/sec
Arm/Group | UroLift
Number analyzed (Participants) | 12
mL/sec | 14.0 (8.4)

2. Primary Outcome: Pdet at Qmax Assessed Using Urodynamic Testing (Cystometry)
Description: Pdet is detrusor pressure at Qmax (maximum urinary flow rate) measured in cm H2O.
Time Frame: 3 Month
Population: Overall number of participants analyzed is fewer than the total number of participants (12) and number of participants analyzed at baseline (8) because unable to interpret data collected at 3 months.
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | UroLift
Number analyzed (Participants) | 8
cm H2O | 82.4 (21.9)

3. Primary Outcome: Pdetmax Assessed Using Urodynamic Testing (Cystometry)
Description: Pdetmax is the maximum void pressure measured in cm H2O.
Time Frame: 3 Month
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | UroLift
Number analyzed (Participants) | 8
cm H2O | 101.5 (30.7)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 1 day, until the AE was resolved, during the 1-3 Day Visit after release from procedure time frame.
Description: Not applicable - Adverse event and/or serious adverse event definition used in this study is the same as defined on clinicaltrials.gov.
Arm/Group | UroLift
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UroLift (N=12)
Urinary retention (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agree not to make any Publications of Study results until completion of the Study and Publication of the results in a peer-reviewed journal by Sponsor. Thereafter, PI may publish their individual site experience. Should a manuscript not be submitted by Sponsor within 12 months of study closure, PI may publish study results. PI shall provide Sponsor 30 days prior notice of publication submission date and text of proposed Publication for review.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/20/NCT04271020/Prot_SAP_000.pdf